CLINICAL TRIAL: NCT05104450
Title: Pragmatic Obstructive Sleep Apnea Weight Loss Trial Assessing Effectiveness and Reach (POWER)
Brief Title: Pragmatic Obstructive Sleep Apnea Weight Loss Trial Assessing Effectiveness and Reach
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 20-240; I01HX003319 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-03 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Sleep Apnea, Obstructive
Keywords: weight loss; lifestyle; diet; exercise; randomized controlled trial
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign participants to one of two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lifestyle intervention (Experimental): The investigators will provide participants with the behavioral lifestyle intervention in addition to usual care.
  Interventions: Behavioral: lifestyle intervention
- usual care control (No Intervention): Participants in this arm will continue with usual care without the lifestyle intervention.

INTERVENTIONS:
Behavioral: lifestyle intervention — Intervention Arm: Usual Care plus a lifestyle behavior change intervention aimed at improving eating habits and increasing physical activity. The lifestyle behavior change intervention encourages participants to gradually achieve and maintain a 5-10% loss of baseline body weight and at least 150 minutes of moderate-intensity physical activity, such as brisk walking, each week. The lifestyle intervention program consists of watching one video, completing corresponding written self-guided learning materials, and tracking food intake and physical activity each week for the first 12 weeks, then working through 10 additional written handouts and continued food and activity tracking for the next nine months. Intervention participants will have access to a lifestyle coach as desired for the full 12-month intervention period.
  Arms: lifestyle intervention

SUMMARY:
Prevalent obesity related conditions like obstructive sleep apnea (OSA) represent an important opportunity to improve population health. OSA reduces quality of life and is associated with greater risk for cardiovascular disease. Although obesity is the single greatest reversible risk factor for OSA, patients with OSA and obesity rarely receive weight loss care to reverse OSA and other serious comorbidities. Efficacy trials reinforce that time and resource intensive lifestyle-based weight loss programs improve weight and physiologic measures of OSA severity (apnea hypopnea index, AHI). However, there are barriers to translating these findings into meaningful gains for population health. To meet these challenges, the investigators propose a pragmatic trial of proactively offering a remote video-based and self-directed lifestyle-based weight loss intervention with remote coaching to patients with OSA. The investigators primary aim is to test the effectiveness of a proactively delivered and pragmatic lifestyle intervention to improve co-primary endpoints of sleep-related quality of life and weight among patients with OSA and obesity. Secondarily, the investigators will compare additional outcomes between groups including cardiovascular risk scores, sleep symptoms, AHI, well-being, and global ratings of change. Finally, the investigators will also conduct an implementation process evaluation informed by the RE-AIM framework to identify barriers and facilitators to widespread implementation.

The investigators will identify patients with OSA and obesity nationwide (n=696) in VA using data from the VA's Corporate Data Warehouse (CDW), and the investigators will contact potentially eligible patients. After confirming eligibility and consent, the investigators will randomly assign subjects to receive the study's lifestyle intervention or usual care alone. The study uses CDW to assess weight change. Subjects will complete questionnaires at baseline at 3, 12 and 21 months after randomization. The lifestyle intervention in POWER focuses on gradual lifestyle behavior change aimed at improving eating habits and increasing physical activity. It encourages participants to gradually achieve and maintain a 5-10% loss of baseline body weight and at least 150 minutes of moderate-intensity physical activity, such as brisk walking, each week. The lifestyle intervention program consists of watching one video, completing corresponding written self-guided learning materials, and tracking food intake and physical activity each week for the first 12 weeks, then working through 10 additional written handouts and continued food and activity tracking for the next nine months. Intervention participants will have access to a lifestyle coach as desired for the full 12-month intervention period.

DETAILED DESCRIPTION:
1. Objective(s) and Hypotheses:

   The investigators' primary aim is to test the effectiveness of a proactively delivered and pragmatic weight loss intervention to improve co-primary endpoints of sleep-related quality of life and weight among Veterans with obstructive sleep apnea (OSA) and obesity.

   Secondarily, the investigators will compare additional outcomes between groups including cardiovascular risk scores, sleep symptoms, AHI, well-being, and global ratings of change. The investigators will also conduct an implementation process evaluation informed by the RE-AIM framework to identify predictors and determinants of population uptake of the intervention.
2. Research Design:

   The investigators plan a hybrid type 1 pragmatic randomized controlled trial assessing effectiveness and an implementation process evaluation.
3. Methodology The investigators will proactively identify patients with OSA and obesity nationwide in VA using data from the CDW (n=696), randomizing patients 1:1 to usual care plus the lifestyle-based weight loss intervention or usual care alone. The investigators will collect primary outcomes at 12 months, but will also collect outcomes at 3 and up to 21 months to assess trends over time.
4. Findings/Progress to Date:

Recruitment and outcome collection completed, analysis is ongoing and not yet complete.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obstructive sleep apnea (OSA) on sleep study (sleep provider confirmed)
* Recent body mass index between 30.0-44.9 kg/m2 and at least one additional plausible BMI in last 12 months
* Access to DVD player, computer, and/or internet
* Able to participate fully in all study protocol/procedures including informed consent

Exclusion Criteria:

* Inability to speak, read, or understand English
* Recent or active weight loss interventions including use of prescription weight-loss medications, participation in group or individual weight loss programs provided by trained personnel, and prior bariatric surgery or plans for bariatric surgery during the study period.
* Expected weight loss because of alternate explanations such as from illness
* High variability in weight due to fluctuations in volume status (e.g. ascites - liver disease, chronic heart failure)
* Safety and/or adherence concerns due to severe physical or mental health issues, or life expectancy <24 months
* Pregnant, lactating, or planning to become pregnant during the study period
* Participation in other intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas M Donovan, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Intervention: The investigators will provide participants with the behavioral lifestyle intervention in addition to usual care.
  The lifestyle behavior change intervention is aimed at improving eating habits and increasing physical activity. The lifestyle behavior change intervention encourages participants to gradually achieve and maintain a 5-10% loss of baseline body weight and at least 150 minutes of moderate-intensity physical activity, such as brisk walking, each week. The lifestyle intervention program consists of watching one video, completing corresponding written self-guided learning materials, and tracking food intake and physical activity each week for the first 12 weeks, then working through 10 additional written handouts and continued food and activity tracking for the next nine months. Intervention participants will have access to a lifestyle coach as desired for the full 12-month intervention period.
Period: Overall Study
Arm/Group | Lifestyle Intervention | Usual Care Control
Started | 348 | 348
Completed | 344 | 345
Not Completed | 4 | 3
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Usual Care Control | Total
Number analyzed (Participants) | 348 | 348 | 696
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.03 (12.03) | 56.38 (12.38) | 56.20 (12.20)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender, Self-Report: Women | 76 | 61 | 137
  Gender, Self-Report: Men | 271 | 285 | 556
  Gender, Self-Report: Non-binary | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 46 | 85
  Not Hispanic or Latino | 308 | 302 | 610
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 55 | 120
  White | 232 | 255 | 487
  More than one race | 29 | 23 | 52
  Unknown or Not Reported | 13 | 11 | 24
OSA Severity [Count of Participants; unit: Participants] — Using sleep studies performed in usual care, we classified individuals as having either mild or moderate-to-severe obstructive sleep apnea (OSA) based on the documented clinical interpretation of the interpreting physician. If the physician did not describe severity in their impression, we classified individuals with an apnea hypopnea index ≥15 events/hour as being moderate-to-severe and all others as mild.
  Participants
    OSA Severity-mild | 116 | 119 | 235
    OSA Severity-moderate to severe | 232 | 229 | 461
BMI [Count of Participants; unit: Participants] — BMI (Body Mass Index) defined based on clinical weight and height. We classified individuals into categories defined by 30-34.9 vs. 35-44.9 kg/m2.
  Participants
    BMI 30-34.9 | 186 | 181 | 367
    BMI 35-44.9 | 162 | 167 | 329
Sleep-related impairment t-score <60 [Count of Participants; unit: Participants] — Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment T-score. Individuals' responses are used to generate a T-score, corresponding to a population mean of 50 with standard deviation of 10. We classified individuals based on T-score values of ≥ 60 vs. <60. A higher PROMIS T-score represents greater Sleep Related Impairment.
  Participants
    Sleep-related impairment t-score <60 | 162 | 161 | 323
    Sleep-related impairment t-score >=60 | 186 | 187 | 373
Charlson Co-Morbidity Index [Mean (Standard Deviation); unit: units on a scale] — Charlson Comorbidity Index (CCI). Individuals receive a score based on their diagnosed comorbidities. These scores range from 0-29. Higher scores indicate a greater mortality risk.
  units on a scale | 0.76 (1.49) | 0.82 (1.45) | 0.79 (1.47)
Rurality/Nonmetropolitan [Count of Participants; unit: Participants] | 52 | 55 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep-related Quality of Life
Description: The investigators will compare change in Functional Outcomes of Sleep questionnaire (FOSQ) score between groups.
  The minimum value of FOSQ is 5, the maximum is 20, and a higher value indicates a better outcome.
Time Frame: baseline to 12 months post randomization
Population: The investigators report here the unadjusted mean changes between baseline and 12 month follow-up. The analysis population for adjusted between-group differences includes participants with a measurement at baseline and/or 12 month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 272 | 315
units on a scale | 1.43 (2.73) | 0.93 (2.89)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; Linear mixed effects model including baseline and follow up outcome measures, time, treatment by time interaction, baseline covariates: age, gender, race, charlson comorbidity index, rurality, and randomization stratification variables: BMI (30-34.9 vs. 35-44.9kg/m2), OSA severity (mild vs. moderate to severe), and sleep related impairment T-score (<60 vs. ≥ 60). The parameter of interest is treatment by time interaction coefficient, measuring the between group difference for change in outcome; Test type: Superiority; p = 0.001, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.64, 95% CI 2-sided [0.25 to 1.04] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

2. Primary Outcome: Change in Weight
Description: The investigators will compare change in weights between intervention and control using clinic weights from VA medical record
Time Frame: baseline to between 9 and 15 months post randomization
Population: The investigators report here the unadjusted mean changes between baseline and 9-to-15 month post-randomization follow-up. The analysis population for adjusted between-group differences includes participants with a measurement at baseline and/or 9-to-15 month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 285 | 291
kg | -2.10 (6.75) | -0.88 (5.86)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.037, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -1.06, 95% CI 2-sided [-2.05 to -0.06] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

3. Secondary Outcome: Cardiovascular Risk Scores
Description: The investigators will compare change in cardiovascular risk scores between intervention and control using the non-laboratory Framingham algorithm. The minimum value in this risk score is -2, the maximum is 32, and a higher value indicates greater risk of cardiovascular disease (worse outcome).
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 346 | 347
score on a scale | 0.22 (3.47) | -0.20 (3.65)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.135, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.37, 95% CI 2-sided [-0.12 to 0.86] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

4. Secondary Outcome: PROMIS - Sleep Disturbance Survey Change
Description: The investigators will compare change in sleep disturbance between intervention and control using the Patient Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Survey. Individuals' responses are used to generate a T-score, corresponding to a population mean of 50 with standard deviation of 10. The minimum value for PROMIS Sleep Disturbance is a T-score of 28.9, the maximum is a T-score of 76.5, and a greater value indicates greater sleep disturbance (worse outcome).
Time Frame: baseline to 3 months post randomization
Population: The investigators report here the unadjusted mean changes between baseline and 3 month follow-up. The analysis population for adjusted between-group differences includes participants with a measurement at baseline and/or 3 month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 241 | 304
T-score | -3.34 (7.69) | -3.02 (6.76)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.068, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -0.97, 95% CI 2-sided [-2.01 to 0.07] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

5. Secondary Outcome: PROMIS - Sleep Related Impairment Survey Change
Description: The investigators will compare change in sleep-related impairment between intervention and control using the Patient Reported Outcomes Measurement Information System (PROMIS) -Sleep Related Impairment Survey. Individuals' responses are used to generate a T-score, corresponding to a population mean of 50 with standard deviation of 10. The minimum value for PROMIS Sleep Related Impairment is a T-score of 30.0, the maximum is a T-score of 80.1, and a greater value indicates greater sleep related impairment (worse outcome).
Time Frame: baseline to 3 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 242 | 306
T-score | -5.67 (8.84) | -3.13 (7.76)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -2.71, 95% CI 2-sided [-3.83 to -1.60] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

6. Secondary Outcome: Systolic Blood Pressure From VA Medical Record
Description: The investigators will compare change in systolic blood pressure values between intervention and control.
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 291 | 295
millimeters of mercury (mm Hg) | -0.22 (15.73) | -2.26 (15.06)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.401, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.87, 95% CI 2-sided [-1.16 to 2.89] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

7. Secondary Outcome: Treatment Usage Per Day
Description: The investigators will compare change in daily OSA treatment usage between groups using self-report.
Time Frame: baseline to 3 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 239 | 300
hours per night | 1.04 (2.99) | 1.58 (3.48)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.034, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -0.51, 95% CI 2-sided [-0.98 to -0.04] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

8. Secondary Outcome: Apnea Hypopnea Index 1b Criteria
Description: The investigators will conduct home sleep apnea tests among a subset of patients in each group to compare apnea hypopnea index (a physiologic measure of OSA severity) between groups at 12 months. The apnea hypopnea index measures the number of times per hour of sleep in which an individual stops breathing (apnea) or nearly stops breathing (hypopnea). For this outcome, we will measure apneas and hypopneas using the 1B criteria of the American Academy of Sleep Medicine.
Time Frame: 12 months post randomization
Population: The investigators report here the unadjusted means for this outcome. The analysis population for adjusted between-group differences includes participants with available covariate data; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 79 | 103
events per hour | 13.77 (14.53) | 16.49 (17.73)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; Linear mixed effects model including each participant's outcome measure, baseline covariates: age, gender, race, charlson comorbidity index, rurality, and randomization stratification variables: BMI (30-34.9 vs. 35-44.9kg/m2), OSA severity (mild vs. moderate to severe), and sleep related impairment T-score (<60 vs. ≥ 60); Test type: Superiority; p = 0.061, Mixed Models Analysis; one-time measures: Beta Estimates; Mean Difference (Final Values) = -3.11, 95% CI 2-sided [-6.37 to 0.15] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

9. Secondary Outcome: Longer-term Change in Weight
Description: The investigators will compare longer-term change in weight between intervention and control using clinic weights from VA medical record
Time Frame: baseline to between 18 and 24 months post randomization
Population: The investigators report here the unadjusted mean changes between baseline and 18-to-24 month post-randomization follow-up. The analysis population for adjusted between-group differences includes participants with a measurement at baseline and/or 18-to-24 month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 260 | 274
kg | -2.64 (7.71) | -1.98 (7.79)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.469, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -0.46, 95% CI 2-sided [-1.69 to 0.78] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

10. Secondary Outcome: Short-term Change in Sleep-related Quality of Life
Description: The investigators will compare short-term change in Functional Outcomes of Sleep questionnaire (FOSQ) between groups. The minimum value of FOSQ is 5, the maximum is 20, and a higher value indicates a better outcome.
Time Frame: baseline to 3 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 247 | 310
units on a scale | 1.30 (2.34) | 0.67 (2.35)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.78, 95% CI 2-sided [0.42 to 1.13]; Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

11. Secondary Outcome: Longer-term Change in Sleep-related Quality of Life
Description: The investigators will compare longer-term change in Functional Outcomes of Sleep questionnaire (FOSQ) between groups. The minimum value of FOSQ is 5, the maximum is 20, and a higher value indicates a better outcome.
Time Frame: baseline to 21 months post randomization
Population: The investigators report here the unadjusted mean changes between baseline and 21 month follow-up. The analysis population for adjusted between-group differences includes participants with a measurement at baseline and/or 21 month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 249 | 302
units on a scale | 1.29 (3.08) | 0.96 (2.89)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.031, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.47, 95% CI 2-sided [0.04 to 0.89] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

12. Secondary Outcome: Global Rating of Change
Description: The investigators will compare perceived change in symptoms between groups using the single-item patients' global impression of change (PGI-C). PGI-C has been validated in the context of OSA treatment and asks patients to rate symptom changes on a 7 point scale from "1-Very Much Improved" to "7-Very Much Worse".
Time Frame: 3 months post randomization
Population: The investigators report here the unadjusted means for this outcome at 3-month follow-up. The analysis population for adjusted between-group differences includes participants with available covariate data; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 240 | 300
units on a scale | 3.29 (1.00) | 3.40 (1.00)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.118, Mixed Models Analysis; one-time measures: Beta Estimates; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.21 to 0.02] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

13. Secondary Outcome: Change in Self-reported Well-being
Description: The investigators will compare change in self-reported well-being between groups. Participants will complete a 3-item Well-being signs (WBS) survey asking them to rate the proportion of time they are satisfied, involved, and functioning their best in activities that they value. The minimum value is 0% and the maximum value is 100%, and a higher value on WBS indicates a better outcome.
Time Frame: baseline to 3 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 240 | 302
units on a scale | 7.76 (20.92) | 3.54 (19.63)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 3.93, 95% CI 2-sided [0.91 to 6.95] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

14. Secondary Outcome: Cardiovascular Risk Scores
Description: The investigators will compare cardiovascular risk scores between intervention and control using the non-laboratory Framingham algorithm. The minimum value in this risk score is -2, the maximum is 32, and a higher value indicates greater risk of cardiovascular disease (worse outcome).
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 344 | 345
score on a scale | 0.35 (3.49) | -0.14 (3.51)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.074, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.44, 95% CI 2-sided [-0.04 to 0.93] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

15. Secondary Outcome: PROMIS - Sleep Disturbance Survey Change
Description: The investigators will compare sleep-related disturbance between intervention and control using the Patient Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Survey.
  Individuals' responses are used to generate a T-score, corresponding to a population mean of 50 with standard deviation of 10. The minimum value for PROMIS Sleep Disturbance is a T-score of 28.9, the maximum is a T-score of 76.5, and a greater value indicates greater sleep disturbance (worse outcome).
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 263 | 301
T-score | -4.53 (8.08) | -3.21 (8.01)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -1.71, 95% CI 2-sided [-2.82 to -0.59] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

16. Secondary Outcome: PROMIS - Sleep Disturbance Survey Change
Description: as for outcome 15
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 238 | 293
T-score | -3.88 (7.75) | -3.44 (8.32)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.229, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -0.70, 95% CI 2-sided [-1.84 to 0.44] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

17. Secondary Outcome: PROMIS - Sleep Related Impairment Survey Change
Description: The investigators will compare sleep-related impairment between intervention and control using the Patient Reported Outcomes Measurement Information System (PROMIS) -Sleep Related Impairment Survey. Individuals' responses are used to generate a T-score, corresponding to a population mean of 50 with standard deviation of 10. The minimum value for PROMIS Sleep Related Impairment is a T-score of 30.0, the maximum is a T-score of 80.1, and a greater value indicates greater sleep related impairment (worse outcome).
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 263 | 303
T-score | -6.33 (9.04) | -3.96 (9.79)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -2.51, 95% CI 2-sided [-3.72 to -1.29] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

18. Secondary Outcome: PROMIS - Sleep Related Impairment Survey Change
Description: as for outcome 17
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 238 | 294
T-score | -5.78 (9.78) | -4.76 (9.88)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.116, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = -1.02, 95% CI 2-sided [-2.30 to 0.25] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

19. Secondary Outcome: Systolic Blood Pressure From VA Medical Record
Description: The investigators will compare change in systolic blood pressure values between intervention and control.
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 210 | 209
millimeters of mercury (mm Hg) | -0.67 (15.20) | -2.25 (15.10)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.968, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.05, 95% CI 2-sided [-2.35 to 2.45] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

20. Secondary Outcome: Diastolic Blood Pressure From VA Medical Record
Description: The investigators will compare change in diastolic blood pressure values between intervention and control.
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 291 | 295
millimeters of mercury (mm Hg) | -0.30 (10.57) | -1.44 (9.78)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.218, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.84, 95% CI 2-sided [-0.49 to 2.17] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

21. Secondary Outcome: Diastolic Blood Pressure From VA Medical Record
Description: The investigators will compare change in diastolic blood pressure values between intervention and control.
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 210 | 209
millimeters of mercury (mmHg) | 0.13 (10.42) | -1.74 (9.54)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.212, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 1.02, 95% CI 2-sided [-0.58 to 2.62] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

22. Secondary Outcome: Treatment Usage Per Day
Description: The investigators will compare change in daily OSA treatment usage between groups using self-report.
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours of use
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 259 | 303
hours of use | 1.45 (3.68) | 1.43 (3.78)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.800, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.44 to 0.57] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

23. Secondary Outcome: Treatment Usage Per Day
Description: The investigators will compare change in daily OSA treatment usage between groups using self-report.
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours of usage
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 235 | 290
hours of usage | 1.47 (3.71) | 1.23 (3.95)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.317, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.26 to 0.79] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

24. Secondary Outcome: Global Rating of Change
Description: as for outcome 12
Time Frame: 12 months post randomization
Population: The investigators report here the unadjusted means for this outcome at 12-month follow-up. The analysis population for adjusted between-group differences includes participants with available covariate data; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 262 | 304
units on a scale | 3.05 (1.15) | 3.25 (1.20)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; one-time measures: Beta Estimates; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.44 to -0.17] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

25. Secondary Outcome: Global Rating of Change
Description: as for outcome 12
Time Frame: 21 months post randomization
Population: The investigators report here the unadjusted means for this outcome at 21-month follow-up. The analysis population for adjusted between-group differences includes participants with available covariate data; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 233 | 293
units on a scale | 2.91 (1.21) | 3.10 (1.23)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.107, Mixed Models Analysis; one-time measures: Beta Estimates; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.27 to 0.03] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

26. Secondary Outcome: Change in Self-reported Well-being
Description: as for outcome 13
Time Frame: baseline to 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 263 | 303
units on a scale | 9.70 (20.73) | 5.50 (24.14)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.013, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 4.07, 95% CI 2-sided [0.86 to 7.27] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

27. Secondary Outcome: Change in Self-reported Well-being
Description: as for outcome 13
Time Frame: baseline to 21 months post randomization
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 234 | 293
units on a scale | 7.96 (21.68) | 5.24 (23.07)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.065, Mixed Models Analysis; treatment-by-time interaction; Mean Difference (Net) = 3.11, 95% CI 2-sided [-0.20 to 6.42] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

28. Secondary Outcome: Apnea Hypopnea Index 1a Criteria
Description: The investigators will conduct home sleep apnea tests among a subset of patients in each group to compare apnea hypopnea index (a physiologic measure of OSA severity) between groups at 12 months. The apnea hypopnea index measures the number of times per hour of sleep in which an individual stops breathing (apnea) or nearly stops breathing (hypopnea). For this outcome, we will measure apneas and hypopneas using the 1A criteria of the American Academy of Sleep Medicine.
Time Frame: 12 months post randomization
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 79 | 103
events per hour | 20.06 (16.05) | 23.23 (19.18)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.041, Mixed Models Analysis; one-time measures: Beta Estimates; Mean Difference (Final Values) = -3.63, 95% CI 2-sided [-7.11 to -0.14] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

ADVERSE EVENTS:
Time Frame: We systematically collected adverse events (AE) by body system as part of the the 12- and 21-month follow-up survey process. For conditions that participants indicated were new since their baseline visit, study staff conducted electronic health record chart review for details of that condition. We also systematically reviewed the electronic health record for discharge summaries among all participants at 12 months, and at 21 month follow-up among those who did not complete follow-up surveys.
Description: Adverse Events were monitored/assessed without regard to specific Adverse Event Terms.
Arm/Group | Lifestyle Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 1/348 | 2/348
Serious Adverse Events (participants affected / at risk) | 54/348 | 40/348
Other Adverse Events (participants affected / at risk) | 126/348 | 127/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lifestyle Intervention (N=348) | Usual Care Control (N=348)
Hematological (Blood and lymphatic system disorders) | 5 | 4
Cardiovascular (Cardiac disorders) | 17 | 21
Gastrointestinal (Gastrointestinal disorders) | 10 | 6
Other (General disorders) | 5 | 2
Hepatobiliary (Hepatobiliary disorders) | 3 | 0
Metabolic (Metabolism and nutrition disorders) | 2 | 3
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 | 7
Neurological (Nervous system disorders) | 9 | 2
Psychological (Psychiatric disorders) | 4 | 3
Renal/Urologic (Renal and urinary disorders) | 6 | 5
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dermatological (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lifestyle Intervention (N=348) | Usual Care Control (N=348)
Hematological (Blood and lymphatic system disorders) | 1 | 1
Cardiovascular (Cardiac disorders) | 21 | 13
Gastrointestinal (Gastrointestinal disorders) | 21 | 21
Other (General disorders) | 21 | 18
Hepatobiliary (Hepatobiliary disorders) | 2 | 3
Metabolic (Metabolism and nutrition disorders) | 4 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 63 | 54
Neurological (Nervous system disorders) | 13 | 12
Psychological (Psychiatric disorders) | 11 | 6
Renal/Urologic (Renal and urinary disorders) | 7 | 15
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 21 | 12
Dermatological (Skin and subcutaneous tissue disorders) | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT05104450/Prot_008.pdf
  • Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT05104450/SAP_006.pdf